CLINICAL TRIAL: NCT05475457
Title: Oregon Supplement: Supporting Sustainable Positive Interactions in the Child Welfare System: The R3 Supervisor Strategy
Status: Completed | Type: Observational
Sponsor: Oregon Social Learning Center (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Other Study IDs: R01DA040416-S1; R01DA040416 (NIH)
Record Dates: First submitted 2022-07-22; First posted 2022-07-27 (Actual); Last update posted 2022-07-27 (Actual); Status verified 2022-07

CONDITIONS: Evidence-Based Practice

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Oregon County 1: First cohort to be trained and monitored with coaching in the R3 model.
  Interventions: Behavioral: R3
- Oregon County 2: Second cohort to be trained and monitored with coaching in the R3 model.
  Interventions: Behavioral: R3

INTERVENTIONS:
Behavioral: R3 — Training, consultation, and fidelity-monitoring to supervisors in the child welfare system to reinforce (1) effort, (2) relationships and roles, and (3) small steps toward goal achievement.

SUMMARY:
This administrative supplement capitalized on the preliminary positive outcomes from the primary parent grant award (R01DA040416), and lessons learned from the implementation of the R3 Supervisor Strategy (R3) throughout the participating four regions (12 counties) in Tennessee. This project aimed to pilot the implementation of R3 with a new sample, a cohort of counties in Oregon particularly affected by the current opioid epidemic, for potential scale-up.

DETAILED DESCRIPTION:
Oregon currently is experiencing a crisis within its Child Welfare System (CWS), with combined challenges within the workforce and departmental support, and a staggering rise in referrals for parental substance abuse. The R3 Supervisor Strategy (R3) provides training, consultation, and fidelity-monitoring to supervisors in the CWS, who are centrally positioned between caseworkers (who have daily interactions with CWS-involved families) and leadership (who make decisions that affect the organization in which families receive services). Supervisors are trained to implement key reinforcement strategies that make up the three Rs including reinforcement of (1) effort, (2) relationships and roles, and (3) small steps toward goal achievement. R3 is relatively easy to learn and sustain and has demonstrated promise in improving CWS outcomes in the parent grant award (R01DA040416). Because many of the counties most impacted by the opioid crisis are rural and under-resourced, an approach like R3 provides the opportunity to introduce evidence-based strategies to these regions where it otherwise is not feasible to adopt more intensive services. This study utilized the same Hybrid Type II design as its parent grant in which supervisors and caseworkers from two Oregon counties particularly affected by the substance abuse crisis were recruited to to provide a pilot assessment of the effectiveness of R3 with an emphasis on referrals for opioid and methamphetamine use (Aim 1). In doing so, the study also sought to modify the R3 training materials to emphasize examples of working with families referred for parental substance abuse (Aim 2) and replicate the preliminary findings from the parent grant, providing pilot data for a larger state scale-up of R3. This administrative supplement allowed an initial assessment to identify if R3's strategies are profound enough to impact the most challenging systems, faced with the most challenging public health crisis presented currently-the impact of the opioid epidemic on families.

ELIGIBILITY:
Inclusion Criteria:

* Oregon Child welfare workforce employee in a participating county.

Exclusion Criteria:

- Contract Workers

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Study participants include casework supervisors in the child welfare system (CWS) from two counties most heavily impacted by the opioid and methamphetamine crisis (Lane and Douglas county).
Sampling Method: Non-Probability Sample
Enrollment: 404 (Actual)
Dates: Start 2019-04-08 (Actual); Primary Completion 2021-07-16 (Actual); Study Completion 2021-07-16 (Actual)

PRIMARY OUTCOMES:
Mean Changes in Organizational Support of Evidence-Based Practices from Baseline to 18-Months Post-Baseline | Baseline to 18-months Post-Baseline
  Changes in overall organizational support of evidence-based practices (i.e., R3) as measured through the Implementation Citizenship Behavior Scale's (ICBS) total score. Measured at Baseline, 6-, 12-, and 18-months Post-Baseline.
Mean Changes in Organizational Assistance Implementing Evidence-Based Practices from Baseline to 18-Months Post-Baseline | Baseline to 18-months Post-Baseline
  Changes in the organization helping others implement Evidence-Based Practices (i.e., R3) as measured through the Implementation Citizenship Behavior Scale's (ICBS) "Helping Other's" subscale. Measured at Baseline, 6-, 12-, and 18-months Post-Baseline.
Mean Changes in the Organization Keeping Others Informed of Evidence-Based Practices Changes and Needs from Baseline to 18-Months Post-Baseline | Baseline to 18-months Post-Baseline
  Changes in the organization keeping others informed of changes and needs in evidence-based practices (i.e., R3) as measured through the Implementation Citizenship Behavior Scale's (ICBS) "Keeping Informed" subscale. Measured at Baseline, 6-, 12-, and 18-months Post-Baseline.
Mean Changes in the Organizational Climate for Implementing Evidence-Based Practices from Baseline to 18-Months Post-Baseline | Baseline to 18-months Post-Baseline
  Changes in organizational climate for implementing evidence-based practices (i.e., R3) as measured by the Implementation Climate Scale's (ICS) total score. Measured at Baseline, 6-, 12-, and 18-months Post-Baseline.
Mean Changes in the Organizational Focus on Evidence-Based Practices from Baseline to 18-Months Post-Baseline | Baseline to 18-months Post-Baseline
  Changes in organizational focus on evidence-based practices (i.e., R3) as measured by the Implementation Climate Scale's (ICS) "Focus on Evidence-Based Practices" subscale. Measured at Baseline, 6-, 12-, and 18-months Post-Baseline.
Mean Changes in the Organization's Educational Support for Evidence-Based Practices from Baseline to 18-Months Post-Baseline | Baseline to 18-months Post-Baseline
  Changes in the organization's educational support for evidence-based practices (i.e., R3) as measured by the Implementation Climate Scale's (ICS) "Educational Support for Evidence-Based Practices" subscale. Measured at Baseline, 6-, 12-, and 18-months Post-Baseline.
Mean Changes in Organizational Recognition for Evidence-Based Practices from Baseline to 18-Months Post-Baseline | Baseline to 18-months Post-Baseline
  Changes in the organization's recognition for evidence-based practices (i.e., R3) as measured by the Implementation Climate Scale's (ICS) "Recognition for Evidence-Based Practices" subscale. Measured at Baseline, 6-, 12-, and 18-months Post-Baseline.
Mean Changes in Organizational Rewards for Evidence-Based Practices from Baseline to 18-Months Post-Baseline | Baseline to 18-months Post-Baseline
  Changes in the organization's rewards for using evidence-based practices (i.e., R3) as measured by the Implementation Climate Scale's (ICS) "Rewards for Evidence-Based Practices" subscale. Measured at Baseline, 6-, 12-, and 18-months Post-Baseline.
Mean Changes in the Organization's Selection for Evidence-Based Practices from Baseline to 18-Months Post-Baseline | Baseline to 18-months Post-Baseline
  Changes in the organization's selection for evidence-based practices (i.e., R3) as measured by the Implementation Climate Scale's (ICS) "Selection for Evidence-Based Practices" subscale. Measured at Baseline, 6-, 12-, and 18-months Post-Baseline.
Mean Changes in the Organization's Selection for Openness to New Practices from Baseline to 18-Months Post-Baseline | Baseline to 18-months Post-Baseline
  Changes in the organization's selection for openness to implement new practices as measured by the Implementation Climate Scale's (ICS) "Selection for Openness" subscale. Measured at Baseline, 6-, 12-, and 18-months Post-Baseline.
Mean Changes in Supervisors' Self-Reported Leadership Abilities for Implementation from Baseline to 18-Months Post-Baseline | Baseline to 18-months Post-Baseline
  Changes in supervisors' self-reported leadership abilities for implementing evidence-based practices (i.e., R3) as measured by the Implementation Leadership Scale's (ILS) total score. Measured at Baseline, 6-, 12-, and 18-months Post-Baseline.
Mean Changes in Supervisors' Self-Reported Ability to Provide Proactive Leadership from Baseline to 18-Months Post-Baseline | Baseline to 18-months Post-Baseline
  Changes in supervisors' self-reported ability to provide proactive leadership when implementing evidence-based practices (i.e., R3) as measured by the Implementation Leadership Scale's (ILS) "Proactive Leadership" subscale. Measured at Baseline, 6-, 12-, and 18-months Post-Baseline.
Mean Changes in Supervisors' Self-Reported Ability to Provide Knowledgeable Leadership from Baseline to 18-Months Post-Baseline | Baseline to 18-months Post-Baseline
  Changes in supervisors' self-reported ability to provide knowledgeable leadership when implementing evidence-based practices (i.e., R3) as measured by the Implementation Leadership Scale's (ILS) "Knowledgeable Leadership" subscale. Measured at Baseline, 6-, 12-, and 18-months Post-Baseline.
Mean Changes in Supervisors' Self-Reported Ability to Provide Supportive Leadership from Baseline to 18-Months Post-Baseline | Baseline to 18-months Post-Baseline
  Changes in supervisors' self-reported ability to provide supportive leadership when implementing evidence-based practices (i.e., R3) as measured by the Implementation Leadership Scale's (ILS) "Supportive Leadership" subscale. Measured at Baseline, 6-, 12-, and 18-months Post-Baseline.
Mean Changes in Supervisors' Self-Reported Ability to Provide Perseverant Leadership from Baseline to 18-Months Post-Baseline | Baseline to 18-months Post-Baseline
  Changes in supervisors' self-reported ability to provide perseverant leadership when implementing evidence-based practices (i.e., R3) as measured by the Implementation Leadership Scale's (ILS) "Perseverant Leadership" subscale. Measured at Baseline, 6-, 12-, and 18-months Post-Baseline.
Mean Changes in Supervisors' Leadership Ability for Implementation from Baseline to 18-Months Post-Baseline | Baseline to 18-months Post-Baseline
  Changes in staff perceptions of their supervisors' leadership abilities for implementing evidence-based practices (i.e., R3) as measured by the Implementation Leadership Scale's (ILS) total score. Measured at Baseline, 6-, 12-, and 18-months Post-Baseline.
Mean Changes in Supervisors' Ability to Provide Proactive Leadership from Baseline to 18-Months Post-Baseline | Baseline to 18-months Post-Baseline
  Changes in staff perceptions of their supervisors' ability to provide proactive leadership when implementing evidence-based practices (i.e., R3) as measured by the Implementation Leadership Scale's (ILS) "Proactive Leadership" subscale. Measured at Baseline, 6-, 12-, and 18-months Post-Baseline.
Mean Changes in Supervisors' Ability to Provide Knowledgeable Leadership from Baseline to 18-Months Post-Baseline | Baseline to 18-months Post-Baseline
  Changes in staff perceptions of their supervisors' ability to provide knowledgeable leadership when implementing evidence-based practices (i.e., R3) as measured by the Implementation Leadership Scale's (ILS) "Knowledgeable Leadership" subscale. Measured at Baseline, 6-, 12-, and 18-months Post-Baseline.
Mean Changes in Supervisors' Ability to Provide Supportive Leadership from Baseline to 18-Months Post-Baseline | Baseline to 18-months Post-Baseline
  Changes in staff perceptions of their supervisors' ability to provide supportive leadership when implementing evidence-based practices (i.e., R3) as measured by the Implementation Leadership Scale's (ILS) "Supportive Leadership" subscale. Measured at Baseline, 6-, 12-, and 18-months Post-Baseline.
Mean Changes in Supervisors' Ability to Provide Perseverant Leadership from Baseline to 18-Months Post-Baseline | Baseline to 18-months Post-Baseline
  Changes in staff perceptions of their supervisors' ability to provide perseverant leadership when implementing evidence-based practices (i.e., R3) as measured by the Implementation Leadership Scale's (ILS) "Perseverant Leadership" subscale. Measured at Baseline, 6-, 12-, and 18-months Post-Baseline.
Mean Changes in Organizational Commitment to Implementing Changes from Baseline to 18-Months Post-Baseline | Baseline to 18-months Post-Baseline
  Changes in staff perceptions of their organization's commitment to implementing changes as measured by the Organizational Readiness for Implementing Change's (ORIC) "Change Commitment" subscale. Measured at Baseline, 6-, 12-, and 18-months Post-Baseline.
Mean Changes in Organizational Effectiveness in Implementing Changes from Baseline to 18-Months Post-Baseline | Baseline to 18-months Post-Baseline
  Changes in staff perceptions of their organization's effectiveness in implementing changes as measured by the Organizational Readiness for Implementing Change's (ORIC) "Change Efficacy" subscale. Measured at Baseline, 6-, 12-, and 18-months Post-Baseline.
Mean Changes in Organizational Readiness to Implement Changes from Baseline to 18-Months Post-Baseline | Baseline to 18-months Post-Baseline
  Changes in staff perceptions of their organization's overall readiness in implementing changes as measured by the Organizational Readiness for Implementing Change's (ORIC) total score. Measured at Baseline, 6-, 12-, and 18-months Post-Baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Saldana, PhD, Principal Investigator — OSLC
Locations (1):
- Oregon Social Learning Center, Eugene, Oregon, United States